CLINICAL TRIAL: NCT00230659
Title: Investigation of Coagulation Parameters in Hereditary Haemorrhagic
Brief Title: Investigation of Coagulation Parameters in Hereditary Haemorrhagic Telangiectasia
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Hammersmith Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IC/CLS6
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma sample aliquots.

GROUPS / COHORTS (2):
- HHT patients: Patients with hereditary haemorrhagic telangiectasia. Blood sample to be taken.
  Interventions: Other: Blood sample to be taken.
- Controls: People without hereditary haemorrhagic telangiectasia. Blood sample to be taken.
  Interventions: Other: Blood sample to be taken.

INTERVENTIONS:
Other: Blood sample to be taken. — Blood sample to be taken.

SUMMARY:
We will address coagulation parameters in hereditary haemorrhagic telangiectasia (HHT) compared to controls.

DETAILED DESCRIPTION:
The inherited disease hereditary haemorrhagic telangiectasia (HHT) causes bleeding from dilated fragile vessels, particularly in the nose and gut. However, many HHT patients develop deep venous thromboses and/or pulmonary embolism, necessitating treatments with anticoagulants that further impair control of their haemorrhagic state. Our initial observations using general coagulation tests suggest that the blood of HHT patients is intrinsically hypercoagulable.

We hypothesize that the genetically-determined abnormality in the blood vessels of HHT patients leads to alteration in the concentrations or activity of one or several of the proteins which affect blood clotting leading to a hypercoagulable state.

We propose to study levels and activity of blood coagulation factors in people with hereditary haemorrhagic telangiectasia and in normal volunteers. This should define the significance and basis for our initial observations, and will have significant implications for the clinical management of HHT patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HHT and normal controls

Exclusion Criteria:

* Previous thrombosis, recent ill health

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 'Patients with HHT' have a clinical diagnosis of hereditary haemorrhagic telangiectasia (HHT)
  'Normal controls' have NO clinical diagnosis of hereditary haemorrhagic telangiectasia (HHT), and are not blood relatives of someone with HHT."
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2004-08; Primary Completion 2007-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Shovlin, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Hammersmith Campus, London, United Kingdom

REFERENCES:
- [Result] Shovlin CL, Sulaiman NL, Govani FS, Jackson JE, Begbie ME. Elevated factor VIII in hereditary haemorrhagic telangiectasia (HHT): association with venous thromboembolism. Thromb Haemost. 2007 Nov;98(5):1031-9. PMID 18000608
- [Result] Livesey JA, Manning RA, Meek JH, Jackson JE, Kulinskaya E, Laffan MA, Shovlin CL. Low serum iron levels are associated with elevated plasma levels of coagulation factor VIII and pulmonary emboli/deep venous thromboses in replicate cohorts of patients with hereditary haemorrhagic telangiectasia. Thorax. 2012 Apr;67(4):328-33. doi: 10.1136/thoraxjnl-2011-201076. Epub 2011 Dec 14. PMID 22169361
- [Result] Shovlin CL, Chamali B, Santhirapala V, Livesey JA, Angus G, Manning R, Laffan MA, Meek J, Tighe HC, Jackson JE. Ischaemic strokes in patients with pulmonary arteriovenous malformations and hereditary hemorrhagic telangiectasia: associations with iron deficiency and platelets. PLoS One. 2014 Feb 19;9(2):e88812. doi: 10.1371/journal.pone.0088812. eCollection 2014. PMID 24586400